CLINICAL TRIAL: NCT02304159
Title: A Randomized Study to Evaluate the Safety and Efficacy of Adding Daclatasvir to the Combination of Sofosbuvir (SOF) and Ribavirin (RBV) for 16 Weeks Versus 24 Weeks in Cirrhotic Subjects With Chronic Hepatitis C Infection Genotype 3
Brief Title: Study to Evaluate the Safety and Efficacy of Daclatasvir/Sofosbuvir/Ribavirin for 16 Versus 24 Weeks for HCV Genotype 3 Cirrhotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tarek I. Hassanein, M.D., FACP, FAG, AGAF (Other)
Responsible Party: Sponsor-Investigator, Tarek I. Hassanein, M.D., FACP, FAG, AGAF, President, Southern California Research Center
Organization: Southern California Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444284
Record Dates: First submitted 2014-11-17; First posted 2014-12-01 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis C; Cirrhosis
Keywords: HCV; Genotype 3; Treatment naive; Treatment experienced
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — daclatasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - 16 weeks (Experimental): Combination of sofosbuvir 400 mg daily, ribavirin 1000-1200 mg daily (weight based) and daclatasvir 60 mg daily for 16 weeks
  Interventions: Drug: daclatasvir; Drug: Sofosbuvir, Sovaldi; Drug: Ribavirin
- Group B - 24 weeks (Active Comparator): Combination of sofosbuvir 400 mg daily, ribavirin 1000-1200 mg daily (weight based) and daclatasvir 60 mg daily for 24 weeks
  Interventions: Drug: daclatasvir; Drug: Sofosbuvir, Sovaldi; Drug: Ribavirin

INTERVENTIONS:
Drug: daclatasvir
  Other Names: DCV, BMS-790052, Daklinza
Drug: Sofosbuvir, Sovaldi
  Other Names: SOF
Drug: Ribavirin
  Other Names: RBV

SUMMARY:
This is a randomized, open label, single center safety and efficacy study. At least 40 cirrhotic subjects with HCV genotype 3 will receive standard of care treatment of sofosbuvir and ribavirin (SOF/RBV) as well as 60 mg daily of Daclatasvir (investigational product). Subjects will be randomized in a 1:1 to receive either:

* Group A: 16 weeks of DCV/SOF/RBV
* Group B: 24 weeks of DCV/SOF/RBV

Subjects will return to the study center at various time points throughout the 16 or 24 weeks of treatment in addition to 12 weeks post taking last dose of study drug to monitor safety and efficacy. These visits will be according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written, informed consent must be available from the subject before any study-specific procedures are performed;
2. Male or female 18-75 years of age;
3. All of the following at least 6 months prior to screening visit:

   * Documented HCV infection based on history of a positive serum anti-HCV antibody test and/or detectable levels of HCV RNA >= 10,000 IU/mL, and
   * Documented HCV genotype 3.
4. Subjects with evidence of cirrhosis defined by either a liver biopsy <= 3 years from screening demonstrating a Metavir Fibrosis Score of F4 (or equivalent); OR Fibroscan® <= 1 year from screening > 12.5 kPa. If a subject is evaluated by more than one testing method, then the liver biopsy results take precedence;
5. Women of childbearing potential (WOCBP) must:

   * have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
   * WOCBP must agree to follow instructions for method(s) of contraception for 7 months post-treatment completion.
   * Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the following duration for 7 months post-treatment completion.
   * Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly.
6. At minimum the subject agrees to the use of two methods of contraception, with at least one method being highly effective as listed below:

Highly Effective Methods of Contraception

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug. WOCBP cannot use hormonal contraception as one of the two methods of contraception because there are no data on the effectiveness of systemic hormonal contraceptives in women taking SOF. However, WOCBP can continue to use hormonal contraceptives, if necessary, in addition to 2 other non-hormonal methods of contraception
* Nonhormonal IUDs, such as ParaGard®
* Tubal Ligation
* Vasectomy
* Complete Abstinence - defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

Less Effective Methods of Contraception

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge
* Male condom without spermicide
* Progestin only pills
* Female condom; A male and female condom must not be used together

Azoospermic males, women who are not of childbearing potential and WOCBP who abstain from heterosexual activity on a continuous basis, are exempt from contraceptive requirements. However, WOCBP who abstain from heterosexual activity on a continuous basis must still undergo pregnancy testing.

Exclusion Criteria:

1. Subjects who lack capacity to consent for themselves;
2. HCV Genotypes other than GT-3 infection; mixed genotype infections are not permitted;
3. Liver histology consistent with any other co-existing cause of chronic liver disease (apart from fatty liver and/or Chronic Hepatitis B Virus);
4. Body Mass Index > 40 at the Screening visit;
5. Any of the following within one month of screening:

   * Uncontrolled diabetes;
   * Unstable or uncontrolled thyroid disease (subjects requiring medication to control their thyroid disease are eligible if all other inclusion/exclusion criteria are met).
6. Any of the following within 6 months of screening visit, any of the following:

   * Decompensated liver disease, esophageal variceal bleeding, or a hepatic mass lesion suspicious for hepatocellular carcinoma (HCC);
   * Subjects who have been treated for HCV infection;
   * History of unstable or deteriorating cardiovascular or cerebrovascular disease;
   * Alcohol and/or drug.
7. QTcF ≥ 500 ms at the baseline visit.
8. Any of the following laboratory abnormalities within 8 weeks of the baseline visit:

   * Hemoglobin <8 g/dL;
   * Absolute neutrophil count <0.50 x 103 cells/μL;
   * Platelet count <25 x 103 cells/μL;
   * Total bilirubin >=3 mg/dL or >=34 mol/L (with the exception of subjects with Gilbert's syndrome);
   * Albumin <2.5g/dL;
   * Creatinine Clearance (CrCl) <=50 mL/min (as estimated by Cockcroft and Gault).
   * Serum ALT >=10 × ULN;
   * Alpha-fetoprotein >200ng/mL.
9. Prior exposure to NS5A inhibitors is prohibited but other classes and pegIFN/RBV are acceptable for treatment-experienced subjects;
10. Use of any prohibited or restricted treatment at least is five half-lives or 14 days (whichever is longer) of the first dose of study drug (refer to section 4.5);
11. History of cancer within 1 year of the screening visit with the exception of localized basal or squamous cell carcinoma;
12. Any gastrointestinal disease or surgical procedure that may impact the absorption of study drug. (Subjects who have had cholecystectomy are permitted to enter the study);
13. Known HIV infection;
14. Confirmed, uncontrolled hypertension (any screening systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg should be excluded);
15. Presence or history of non-HCV chronic liver disease, including autoimmune hepatitis, alpha-1-antitrypsin deficiency, hemochromatosis, Wilson's disease, drug- or toxin-induced liver disease, alcohol-related liver disease, primary biliary cirrhosis and sclerosing cholangitis. Subjects with fatty liver and/or chronic hepatitis B virus in addition to HCV may be considered in the study;
16. Uncontrolled seizures disorder;
17. History of hemoglobinopathies, (e.g., thalassemia, sickle cell anemia, spherocytosis) or other cause of hemolytic anemia, including autoimmune causes;
18. Active disease at screening visit known to cause significant alteration in immunologic function including hematologic malignancy, sarcoidosis or autoimmune disorder (e.g., rheumatoid arthritis, systemic lupus erythematosis, leukemia, lymphoma, autoimmune thyroid disease, scleroderma, unstable psoriasis, and multiple sclerosis);
19. Pregnant or lactating women or women who plan to become pregnant during the study;
20. History of hypersensitivity to drugs with a similar biochemical structure to DCV or SOF or RBV;
21. Any other criteria or known contraindication that would exclude the subject from receiving SOF or RBV (per the local label) or DCV;
22. Inability to tolerate oral medication;
23. Subjects, who in the opinion of the Investigator, are not suitable candidates for enrollment or who would not comply with the requirements of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Southern California Research Center, Coronado, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - 16 Weeks: Combination of sofosbuvir 400 mg daily, ribavirin 1000-1200 mg daily (weight based) and daclatasvir 60 mg daily for 16 weeks
  daclatasvir, Daklinza
  Sofosbuvir, Sovaldi
  Ribavirin
- Group B - 24 Weeks: Combination of sofosbuvir 400 mg daily, ribavirin 1000-1200 mg daily (weight based) and daclatasvir 60 mg daily for 24 weeks
  daclatasvir, Daklinza
  Sofosbuvir, Sovaldi
  Ribavirin
Period: Overall Study
Arm/Group | Group A - 16 Weeks | Group B - 24 Weeks
Started | 21 | 18
Completed | 19 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: A total of 39 participants started treatment with sofosbuvir, ribavirin and daclatasvir. 21 were randomized to Group A (16 weeks of treatment). 18 were randomized to Group B (24 weeks of treatment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - 16 Weeks | Group B - 24 Weeks | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.62 (8.15) | 55.72 (6.32) | 55.13 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 5 | 19
  Not Hispanic or Latino | 7 | 13 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Pre-treatment HCV RNA (viral load) [Mean (Standard Deviation); unit: IU/mL] | 3009718.11 (3750275.88) | 3165043.17 (4871398.73) | 3085281.65 (4271365.19)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: This field states the number of participants who had an adverse event
Time Frame: From baseline (start of study drugs) to last day of taking study drugs; an average of 20 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - 16 Weeks | Group B - 24 Weeks
Number analyzed (Participants) | 21 | 18
Participants | 21 | 18

2. Primary Outcome: Number of Participants With Abnormal Safety Laboratory Tests (ALT and/or Total Bilirubin) That Required Discontinuing Study Drugs
Description: This field states the number of participants who had an abnormal ALT that required discontinuing study drugs and/or abnormal Total Bilirubin that required discontinuing study drugs.
Time Frame: From baseline (start of study drugs) to last day of taking study drugs; an average of 20 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - 16 Weeks | Group B - 24 Weeks
Number analyzed (Participants) | 21 | 18
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Undetectable HCV Virus 12 Weeks After Stopping Study Drugs
Description: Sustained Virologic Response (SVR) defined as undetectable HCV RNA 12 weeks after stopping study drugs.
Time Frame: From baseline (start of study drugs) until 12 weeks after stopping study drugs
Population: The analysis covers only the subjects who reached the 12 weeks after stopping study drugs time point. 19 of 21 participants randomized to Group A reached that timepoint and 16 of 18 participants randomized to Group B reached that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - 16 Weeks | Group B - 24 Weeks
Number analyzed (Participants) | 19 | 16
Participants | 19 | 16

ADVERSE EVENTS:
Time Frame: From start of treatment to 12 weeks after stopping treatment.
Groups:
- Group A - 16 Weeks of Treatment: Combination of sofosbuvir 400 mg daily, ribavirin 1000-1200 mg daily (weight based) and daclatasvir 60 mg daily for 16 weeks
  daclatasvir, Daklinza
  Sofosbuvir, Sovaldi
  Ribavirin
- Group A - 24 Weeks of Treatment: Combination of sofosbuvir 400 mg daily, ribavirin 1000-1200 mg daily (weight based) and daclatasvir 60 mg daily for 24 weeks
  daclatasvir, Daklinza
  Sofosbuvir, Sovaldi
  Ribavirin
Arm/Group | Group A - 16 Weeks of Treatment | Group A - 24 Weeks of Treatment
All-Cause Mortality (participants affected / at risk) | 1/21 | 1/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/18
Other Adverse Events (participants affected / at risk) | 21/21 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - 16 Weeks of Treatment (N=21) | Group A - 24 Weeks of Treatment (N=18)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Violence (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - 16 Weeks of Treatment (N=21) | Group A - 24 Weeks of Treatment (N=18)
Flu-like symptoms (General disorders) | 10 (10) | 9 (9)
Mood Changes (Psychiatric disorders) | 8 (8) | 4 (4)
Fatigue (General disorders) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (4)
Decompensation (Hepatobiliary disorders) | 3 (3) | 5 (5)
Decreased Appetite (General disorders) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Study received IND approval in November 2014. Daclatasvir received initial FDA approval in July 2015. Participants were randomized to receive daclatasvir for either 16 or 24 weeks and were followed per standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02304159/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT02304159/ICF_001.pdf